CLINICAL TRIAL: NCT01807065
Title: Randomized Phase II Trial of Sipuleucel T Immunotherapy Preceded by Sensitizing Radiation Therapy and Sipuleucel-T Alone in Patients With Castrate Resistant Metastatic Prostate Cancer
Brief Title: Sipuleucel-T With or Without Radiation Therapy in Treating Patients With Hormone-Resistant Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12367; NCI-2013-00542 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-03-06; First posted 2013-03-08 (Estimated); Results first posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2019-06

CONDITIONS: Adenocarcinoma of the Prostate; Bone Metastases; Hormone-resistant Prostate Cancer; Recurrent Prostate Cancer; Soft Tissue Metastases; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — sipuleucel-T

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (sipuleucel-T) (Experimental): Patients receive sipuleucel-T IV over 60 minutes days 22, 36, and 50.
  Interventions: Biological: sipuleucel-T; Other: laboratory biomarker analysis
- Arm B (radiation therapy, sipuleucel-T) (Experimental): Patients undergo external beam radiation therapy in weeks 1-2. Patients also receive sipuleucel-T as in Arm A.
  Interventions: Biological: sipuleucel-T; Radiation: external beam radiation therapy; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: sipuleucel-T — Given IV
  Other Names: APC 8015; Provenge
Radiation: external beam radiation therapy — Undergo external beam radiation therapy
  Other Names: EBRT
  Arms: Arm B (radiation therapy, sipuleucel-T)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase II trial studies how well giving sipuleucel-T with or without radiation therapy works in treating patients with hormone-resistant metastatic prostate cancer. Vaccines may help the body build an effective immune response to kill tumor cells. Radiation therapy uses high energy x rays to kill tumor cells. It is not yet known whether giving sipuleucel-T vaccine is more effective with or without radiation therapy in treating prostate cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility, based on percent able or willing to receive all three infusions of sipuleucel-T immunotherapy, when combining sipuleucel-T with radiation therapy to a single site of metastasis delivered one week prior to beginning of sipuleucel-T therapy.

SECONDARY OBJECTIVES:

I. To assess the effect of radiation therapy to single metastasis on immune response (antibody and T-cell proliferation to prostate acid phosphate [PAP] and fusion protein PA2024) generated by sipuleucel-T immunotherapy.

II. To assess the effect of external beam radiotherapy to single metastasis on prostate specific antigen (PSA) response to therapy with sipuleucel-T.

III. To assess the effect of external beam radiotherapy to single metastasis on radiographic response rate to therapy with sipuleucel-T.

IV. To assess the time from the onset of therapy with sipuleucel-T +/- radiation to the need for subsequent therapy for prostate cancer.

V. To assess the toxicity associated with sipuleucel-T +/- radiation.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive sipuleucel-T intravenously (IV) over 60 minutes days 22, 36, and 50.

ARM B: Patients undergo external beam radiation therapy in weeks 1-2. Patients also receive sipuleucel-T as in Arm A.

In both arms, treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up until week 60.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented adenocarcinoma of the prostate
* Life expectancy of >= 6 months, Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Metastatic disease as evidenced by soft tissue and/or bony metastases on baseline bone scan and/or computed tomography (CT) scan or magnetic resonance imaging (MRI) of the abdomen or pelvis
* Castration resistant prostatic adenocarcinoma; subjects must have current or historical evidence of disease progression despite castrated level of testosterone (< 50 ng/dL) achieved by orchiectomy or luteinizing hormone-releasing hormone (LHRH) agonist or antagonist therapy; disease progression has to be demonstrated by PSA progression OR progression of measurable disease OR progression of non-measurable disease as defined below:

  * PSA: Two consecutive rising PSA values, at least 7 days apart
  * Measurable disease: >= 20% increase in the sum of the longest diameters of all measurable lesions or the development of any new lesions; the change will be measured against the best response to castration therapy or against the pre-castration measurements if there was no response
  * Non-measurable disease:

    * Soft tissue disease: The appearance of 1 or more lesions, and/or unequivocal worsening of non-measurable disease when compared to imaging studies acquired during castration therapy or against the pre-castration studies if there was no response
    * Bone disease: Appearance of 2 or more new areas of abnormal uptake on bone scan when compared to imaging studies acquired during castration therapy or against the pre-castration studies if there was no response; increased uptake of pre-existing lesions on bone scan does not constitute progression
* White blood cell (WBC) >= 2,500 cells/uL
* Absolute neutrophil count (ANC) >= 1,000 cells/uL
* Platelet count >= 75,000 cells/uL
* Hemoglobin (HgB) >= 9.0 g/dL
* Creatinine =< 2.5 mg/dL
* Total bilirubin =< 2 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST, serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT, serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN
* Prior chemotherapy with 0-2 regimens is allowed
* Prior radiation therapy to prostate or prostate bed is allowed provided it occurred > 3 months before enrollment to the study

Exclusion Criteria:

* The presence of liver, or known brain metastases, malignant pleural effusions, or malignant ascites
* Moderate or severe symptomatic metastatic disease, defined as a requirement for treatment with opioid analgesics for cancer-related pain within 21 days prior to registration
* Eastern Cooperative Oncology Group (ECOG) performance status > 2
* Treatment with chemotherapy within 3 months of registration
* Treatment with any of the following medications or interventions within 28 days of registration:

  * Systematic corticosteroids; use of inhaled, intranasal, and topical steroids is acceptable
  * Any other systemic therapy for prostate cancer (except for medical castration)
* History of external beam radiation therapy to metastatic sites within 1 year of enrollment to the study
* Participation in any previous study involving sipuleucel-T
* Pathologic long-bone fractures, imminent pathologic long-bone fracture (cortical erosion on radiography > 50%) or spinal cord compression
* Concurrent other malignancy with the exception of:

  * Cutaneous squamous cell and basal carcinomas
  * Adequately treated stage 1-2 malignancy
  * Adequately treated stage 3-4 malignancy that has been in remission for >= 2 years at the time of registration
* A requirement for systemic immunosuppressive therapy for any reason
* Any infection requiring parenteral antibiotic therapy or causing fever (temperature > 100.5 degrees Fahrenheit [F] or 38.1 degrees Celsius [C]) within 1 week prior to registration
* Any medical intervention or other condition which, in the opinion of the principal investigator could compromise adherence with study requirements or otherwise compromise the study's objectives

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-06-07; Primary Completion 2018-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cy Stein, MD, PhD, Principal Investigator — City of Hope Medical Center
Locations (3):
- United States (3):
  - City of Hope Medical Center, Duarte, California
  - South Pasadena Cancer Center, Pasadena, California
  - Huntsman Cancer Institute, Univ. of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Twardowski P, Wong JYC, Pal SK, Maughan BL, Frankel PH, Franklin K, Junqueira M, Prajapati MR, Nachaegari G, Harwood D, Agarwal N. Randomized phase II trial of sipuleucel-T immunotherapy preceded by sensitizing radiation therapy and sipuleucel-T alone in patients with metastatic castrate resistant prostate cancer. Cancer Treat Res Commun. 2019;19:100116. doi: 10.1016/j.ctarc.2018.100116. Epub 2018 Dec 20. PMID 30682445

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Sipuleucel-T): Patients receive sipuleucel-T IV over 60 minutes days 22, 36, and 50. Each dose of sipuleucel-T contains a minimum of 50 million activated CD54+ cells.
  sipuleucel-T: Given IV
  laboratory biomarker analysis: Correlative studies
- Arm B (Radiation Therapy, Sipuleucel-T): Patients undergo external beam radiation therapy in weeks 1-2. Radiation given in 10 fractions of 300cGy for a total dose of 3000cGy. Patients also receive sipuleucel-T as in Arm A.
  sipuleucel-T: Given IV
  external beam radiation therapy: Undergo external beam radiation therapy
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Arm A (Sipuleucel-T) | Arm B (Radiation Therapy, Sipuleucel-T)
Started | 25 | 26
Completed | 24 | 25
Not Completed | 1 | 1
Not completed — Receive no sip-T due to IV access | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Sipuleucel-T) | Arm B (Radiation Therapy, Sipuleucel-T) | Total
Number analyzed (Participants) | 24 | 25 | 49
Age, Continuous [Median (Full Range); unit: years] | 64 [45 to 90] | 67 [54 to 81] | 67 [45 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 24 | 25 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 20 | 20 | 40
  Hispanic | 2 | 2 | 4
  Asian | 0 | 2 | 2
  African American | 2 | 0 | 2
  Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 24 | 25 | 49
Gleason Score [Median (Full Range); unit: Gleason grading] — Gleason Scores range from 2-10. Summing scores (1-5) of common (primary) and second most common (secondary) patterns of cells found in a tissue sample. The higher the Gleason Score, the more likely that the cancer will grow and spread quickly. Scores of 6 or less describe cancer cells that look similar to normal cells and suggest that the cancer is likely to grow slowly. A score of 7 suggests intermediate risk for aggressive cancer. Scores of 8 or higher describe cancers that are likely to spread more rapidly, these cancers are referred to as poorly differentiated or high grade.
  Gleason grading | 8 [6 to 10] | 7 [7 to 9] | 8 [6 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Estimated using the product-limit method of Kaplan and Meier.
  Progression is defined as one or more of the following:
  20% increase in the sum of the longest diameters of target measurable lesions over the smallest sum observed (over baseline if no decrease during therapy) using the same techniques as baseline; unequivocal progression of non-measurable disease in the opinion of the treating physician; appearance of any new lesions; PSA increase of 25% from baseline or nadir and by 2ng/uL or greater at 12 weeks; death due to disease without prior documentation of progression and without symptomatic deterioration.
Time Frame: Until progression or death, Up to 2 years.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Sipuleucel-T) | Arm B (Radiation Therapy, Sipuleucel-T)
Number analyzed (Participants) | 24 | 25
Months | 2.46 [2.17 to 2.66] | 3.65 [2.76 to 4.86]
Statistical Analysis 1: Comparison: Arm A (Sipuleucel-T) vs Arm B (Radiation Therapy, Sipuleucel-T); Test type: Other; p = 0.06, Log Rank

2. Secondary Outcome: Number of Participants With Grade 2 or Above Adverse Events
Description: Number of participants with specified adverse event that is grade 2 or above and related to treatment. Graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.0
Time Frame: Up to 60 weeks
Measure: Number; unit: participants
Arm/Group | Arm A (Sipuleucel-T) | Arm B (Radiation Therapy, Sipuleucel-T)
Number analyzed (Participants) | 24 | 25
participants
  Grade 2 : Chills | 3 | 0
  Grade 2 : Fatigue | 1 | 2
  Grade 2 : Infusion Reaction | 1 | 1
  Grade 2 : Decreased Lymphocyte Count | 1 | 0
  Grade 2 : Nausea | 0 | 1
  Grade 2 : Pain in Extremity | 0 | 1
  Grade 2 : Anemia | 0 | 1
  Grade 2 : Anorexia | 0 | 1
  Grade 2 : Headache | 1 | 1
  Grade 2 : Hypertension | 0 | 3
  Grade 3 : Chills | 0 | 0
  Grade 3 : Fatigue | 0 | 0
  Grade 3 : Infusion Reaction | 0 | 0
  Grade 3 : Decreased Lymphocyte Count | 0 | 0
  Grade 3 : Nausea | 0 | 0
  Grade 3 : Pain in Extremity | 0 | 0
  Grade 3 : Anemia | 0 | 1
  Grade 3 : Anorexia | 0 | 0
  Grade 3 : Headache | 0 | 0
  Grade 3 : Hypertension | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of 1 year and 3 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Arm A (Sipuleucel-T) | Arm B (Radiation Therapy, Sipuleucel-T)
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24
Serious Adverse Events (participants affected / at risk) | 1/25 | 1/24
Other Adverse Events (participants affected / at risk) | 25/25 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Sipuleucel-T) (N=25) | Arm B (Radiation Therapy, Sipuleucel-T) (N=24)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Sipuleucel-T) (N=25) | Arm B (Radiation Therapy, Sipuleucel-T) (N=24)
Anemia (Blood and lymphatic system disorders) | 7 (20) | 11 (34)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (3)
Sinus bradycardia (Cardiac disorders) | 7 (19) | 7 (18)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 0 (0)
Watering eyes (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (4)
Constipation (Gastrointestinal disorders) | 0 (0) | 5 (9)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (3) | 3 (3)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3) | 7 (13)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (5)
Angioectasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
dry heaves (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 9 (17) | 2 (2)
Fatigue (General disorders) | 12 (22) | 10 (19)
Fever (General disorders) | 2 (2) | 1 (1)
Flu like symptoms (General disorders) | 1 (1) | 2 (2)
Infusion related reaction (General disorders) | 2 (2) | 2 (3)
Pain (General disorders) | 3 (4) | 4 (9)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1)
apheresis line infection (Infections and infestations) | 0 (0) | 2 (4)
Bruising (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 4 (10)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (2) | 1 (1)
Alkaline phosphatase increased (Investigations) | 4 (11) | 7 (15)
Aspartate aminotransferase increased (Investigations) | 3 (5) | 4 (7)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (2)
Creatinine increased (Investigations) | 2 (3) | 2 (6)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (3)
Neutrophil count decreased (Investigations) | 2 (5) | 1 (2)
Platelet count decreased (Investigations) | 3 (5) | 7 (20)
Weight loss (Investigations) | 1 (3) | 1 (1)
White blood cell decreased (Investigations) | 4 (7) | 3 (7)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 4 (7)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (4)
Hypernatremia (Metabolism and nutrition disorders) | 4 (5) | 2 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 1 (4)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 4 (9)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2) | 2 (6)
Obesity (Metabolism and nutrition disorders) | 1 (2) | 1 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 6 (9)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (5) | 6 (10)
neck stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
enlarged thryroid nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
skin lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (3)
skin lesion - neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (4) | 2 (2)
Facial muscle weakness (Nervous system disorders) | 0 (0) | 2 (6)
Headache (Nervous system disorders) | 3 (5) | 2 (5)
Paresthesia (Nervous system disorders) | 1 (4) | 3 (7)
Radiculitis (Nervous system disorders) | 0 (0) | 1 (1)
Tingling face, hands, and feet (Nervous system disorders) | 1 (1) | 0 (0)
generalized numbness and tingling during (Nervous system disorders) | 1 (1) | 0 (0)
numbness and tingling in right hand (Nervous system disorders) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 2 (4)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 0 (0)
decreased force of urinary stream (Renal and urinary disorders) | 0 (0) | 1 (3)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
'mild skin irritation in the posterior r (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (4)
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
contact dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 11 (33) | 12 (35)
Hypotension (Vascular disorders) | 2 (4) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/65/NCT01807065/Prot_SAP_000.pdf